CLINICAL TRIAL: NCT07124013
Title: An Open-Label, Phase 1 Study to Investigate the Comparability of the Pharmacokinetics of Olomorasib (LY3537982) Between Two Capsule Formulations and to Evaluate the Food Effect in Healthy Japanese Participants
Brief Title: A Study of Olomorasib (LY3537982) in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27293; J3M-JE-JZQL (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-13; First posted 2025-08-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Olomorasib Test (Part A) (Experimental): Olomorasib test formulation administered orally with or without food.
  Interventions: Drug: Olomorasib
- Olomorasib Reference (Part B) (Experimental): Olomorasib reference formulation administered orally with or without food.
  Interventions: Drug: Olomorasib
- Olomorasib Test (Part B) (Experimental): Olomorasib test formulation administered orally with or without food.
  Interventions: Drug: Olomorasib

INTERVENTIONS:
Drug: Olomorasib — Administered orally
  Other Names: LY3537982

SUMMARY:
The purpose of this study is to compare and see how food affects the amount of olomorasib in the blood when olomorasib is taken in two different capsule forms. Participation in the study will last approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants who are overtly healthy as determined by medical evaluation including medical history, 12 lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations.
* Have a body mass index within the range 18.5 to 30.0 kilograms per square meter (kg/m²), inclusive, at screening.
* Participants assigned male at birth (AMAB) may participate in this study.

Exclusion Criteria:

* Have a history of malignancy within 5 years prior to screening except for basal cell or squamous epithelial carcinomas of the skin or in situ carcinoma of the cervix that have been resected with no evidence of metastatic disease for 3 years.
* Have known allergies to olomorasib or any component of the formulation, or related compounds.
* Use of any other investigational drug or device within 30 days or 5 half-lives (if known), whichever is longer, of the first dose of study drug.
* Have previously completed or withdrawn from this study or any other study investigating olomorasib and have previously received olomorasib
* Show evidence of hepatitis B or positive hepatitis B surface antigen.
* Show evidence of hepatitis C or have a positive hepatitis C virus antibody test.
* Show evidence of HIV infection or positive HIV antigen or HIV antibodies.
* Show evidence of syphilis or have a positive syphilis test.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Olomorasib | Day 1 (Predose) through Day 7 (72 Hours Postdose)
PK: Area under the Concentration versus Time Curve from Time Zero to Time t (AUC[0-tlast]) of Olomorasib | Day 1 (Predose) through Day 7 (72 Hours Postdose)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No